CLINICAL TRIAL: NCT01893658
Title: Xolair (Omalizumab) for Treatment of Drug-induced Acute Tubulointerstitial Nephritis (AIN)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients with a condition of interest that resulted in failure to recruit
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Vesna D. Garovic, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-006797
Record Dates: First submitted 2013-06-12; First posted 2013-07-09 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Acute Interstitial Nephritis
Keywords: Interstitial Nephritis; Nephritis; Tubulointerstitial; Renal disease; Kidney
MeSH Terms: conditions — Acute Tubulointerstitial Nephritis; Nephritis, Interstitial; Nephritis; Kidney Diseases | interventions — Omalizumab; Prednisone; Prednisolone

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omalizumab and Prednisone (Active Comparator): Omalizumab in addition to prednisone. Omalizumab will be given once subcutaneously at a dose of 375 mg within 24 hours after receiving prednisone
  Standard clinical therapy with prednisone.
  * Day 1-14: 60 mg/day 14 days (2 weeks)
  * Day 15-28: 40 mg/day (2 weeks)
  * Day 29-35: 30 mg/day (1 week)
  * Day 36-42: 20 mg/day (1 week)
  * Day 43-49: 10 mg/day (1 week)
  * Day 50-56: 5 mg/day (1 week)
  * Subjects will stop taking prednisone on day 57
  If patients weigh less than 60 Kg, the dose will be adjusted accordingly (to equal 1mg/kg/day of prednisone as the starting dose).
  Interventions: Drug: Omalizumab; Drug: Prednisone
- Prednisone (Active Comparator): Standard clinical therapy with prednisone.
  * Day 1-14: 60 mg/day 14 days (2 weeks)
  * Day 15-28: 40 mg/day (2 weeks)
  * Day 29-35: 30 mg/day (1 week)
  * Day 36-42: 20 mg/day (1 week)
  * Day 43-49: 10 mg/day (1 week)
  * Day 50-56: 5 mg/day (1 week)
  * Subjects will stop taking prednisone on day 57
  If patients weigh less than 60 Kg, the dose will be adjusted accordingly (to equal 1mg/kg/day of prednisone as the starting dose).
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Omalizumab — administration of a single dose together with the standard treatment
  Other Names: Xolair
  Arms: Omalizumab and Prednisone
Drug: Prednisone — standard treatment
  Other Names: Prednisolone

SUMMARY:
The investigators goal is to evaluate the role of XOLAIR® in treatment of Acute Tubulointerstitial Nephritis (AIN) with the goal of shortening the duration and dose of prednisone for treatment of drug-induced AIN. Currently there is no good treatment for drug-induced AIN. Prednisone is the standard treatment but is associated with many side-effects when used long-term and at high doses.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects > 18 years old of both genders
2. Biopsy proven acute interstitial nephritis in the native kidneys without evidence of ischemic or glomerular pathology in the biopsy
3. Normal baseline creatinine defined as estimated GFR ≥ 60 ml/min/SA based on MDRD calculation within 1 year prior to renal biopsy
4. Serum creatinine elevation of > 0.3 mg/dL and/or doubling of serum creatinine compared to most recent documented creatinine available (at least within the last year)
5. No immunosuppressants in the last three months including prednisone
6. Women of childbearing potential not using the contraception method can be included as this is a one time dosing and has no known long-term effects.

Exclusion Criteria:

1. Unwillingness to give consent
2. Patients who are Pregnant (positive serum pregnancy test for females) or breast feeding
3. Documented history of an autoimmune disease
4. Inability or unwillingness to take prednisone for the prescribed duration and/or dose
5. Subjects suspected to have non-drug-induced AIN
6. Subjects not meeting the inclusion criteria
7. Subjects with contraindication to administration of omalizumab
8. Prior use of omalizumab
9. Severe hypersensitivity to omalizumab or any component of the product
10. Known elevated IgE level from other disease processes
11. Subjects taking (nonsteroidal antiinflammatory drug) NSAIDs chronically
12. Use of any other investigational agents in the last 30 days
13. Patients with severe medical condition(s) including metastatic cancer, terminal congestive heart failure, severe ischemic heart disease or any other medical condition in which life expectancy is less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Change in serum creatinine | Baseline to three months

SECONDARY OUTCOMES:
Mean individual percentage drop in serum creatinine relative to entry creatinine levels | baseline to 3 months
Percentage of subjects returning to their usual baseline creatinine (+25%) or below | baseline to 3 months
Reduction in Neutrophil gelatinase-associated lipocalcin. | baseline to 3 months
  24 hours, 4 hours, and in 3 months after Xolair treatment
Percentage of subjects requiring renal replacement therapy | baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vesna D. Garovic, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States